CLINICAL TRIAL: NCT00320281
Title: Botulinum Toxin A for the Treatment of Cervical/Shoulder Pain Following Acute Spinal Cord Injury.
Brief Title: Investigating Botulinum Toxin A to Treat Acute Neck/Upper Shoulder Pain Following a New Spinal Cord Injury.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Craig Hospital (Other)
Collaborators: The Craig H. Neilsen Foundation (Other); Allergan (Industry)
Responsible Party: Principal Investigator, Cynthia Harrison-Felix, PhD, Department Director, Craig Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2691
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Results first posted 2013-07-29 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Spinal Cord Injury; Pain
Keywords: Botox
MeSH Terms: conditions — Spinal Cord Injuries; Pain | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): Normal saline injections were used for placebo injections. Injections were based on treatment plan determined in clinical setting by study PI and physical therapist. 25 cc syringe was used and amount of saline injected was unit based on muscles to be injected according to the treatment plan.
  Interventions: Other: placebo
- Botulinum toxin A (Active Comparator): Botulism toxin A dosage was based on plan developed in clinical setting with study PI and physical therapist. Drug was dosed in 25 cc syringe,diluted with normal saline and injections occured based on treatment plan.
  Interventions: Drug: botulinum toxin A

INTERVENTIONS:
Drug: botulinum toxin A — Injection of BTXA into cervical and upper back muscles based on treatment plan prescribed for each participant individually based on muscle soreness and tightness. Injections occured on one single clinic visit.Both the saline and BTXA were dosed in 25 cc syringes and looked the same for the physician performing the injections to ensure both participant and study physician remained blinded.
  Other Names: Botox-A
  Arms: Botulinum toxin A
Other: placebo — Injection of normal saline into cervical and upper back muscles was also based on treatment plan prescribed for each participant individually based on muscle soreness and tightness. Injections occured on one single clinic visit. Both the saline and BTXA were dosed in 25 cc syringes and looked the same for the physician performing the injections to ensure both participant and study physician remained blinded.
  Other Names: normal saline dose based on muscles to be injected, multiple injections may occur based on treatment plan. Injection occur at one single clinical visit.
  Arms: placebo

SUMMARY:
As clinicians, it is often a struggle to find effective pain control for a certain subgroup of patients with tetraplegia. These patients often have severe upper back, neck, and shoulder pain, limiting rehabilitation productivity and potential, and always limiting quality of life.

This pain appears to be primarily musculoskeletal. Muscles in the upper back and neck become shortened, rock hard, and extremely tender with even the slightest touch or stretch. Refractory to multiple classes of medications, modalities, and other treatments, patients truly suffer-not only from pain, but from fatigue, sedation, expense, and loss of useful rehabilitation time due to attempted remedies. Unfortunately, this subgroup of patients is not small and the problem is significant, as anyone who specializes in the treatment of spinal cord injury patients will recognize.

In search for another form of treatment, botulinum toxin A (BTXA) may be promising for pain control in that group of patients with tetraplegia whose pain has proven to be refractory to treatment. It did not take long searching the literature to find compelling evidence that BTXA may have another mechanism of action for direct pain control, apart from its well known mechanism for spasticity control. Clinically, it is increasingly being recommended and used for this purpose. In fact, one of the specific indications now recognized by most for BTXA treatment is for myogenic pain due to short, tight, strained muscles-just as we see with our population. Yet, it's application has not been studied in people with tetraplegia. Thus, the genesis of the project and the hope to help our patients evolved.

Study hypotheses:

* In addition to traditional treatments used for pain control, injection of BTXA into cervical and upper back muscles will effectively reduce cervical/shoulder pain severity reported by individuals with cervical spinal cord injuries, regardless of the etiology of pain.
* Pain reduction secondary to the use of BTXA will be associated with a decrease in total analgesic medication use among SCI patients during acute inpatient rehabilitation.
* BTXA to treat cervical/shoulder pain will increase active participation in the rehabilitation program for individuals with tetraplegia during inpatient rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient at Craig Hospital for initial rehabilitation following a traumatic spinal cord injury.
* Cervical Injury at C4-C8
* ASIA classification score of A,B,or C
* May still be in halo immobilization device and range of motion scores will therefore not be collected
* Report at least a 6/10 on the VAS for pain in the previous 24 hours prior to randomization
* Orthopedically stable
* Approval of attending physician
* Standard of care management with oral analgesic agents has not resulted in pain symptom resolution
* May not be enrolled in other clinical trial

Exclusion Criteria:

* Pregnant
* Concurrent use of aminoglycoside antibiotics at the time of injection
* Diagnosis of myasthenia gravis or Eaton-Lambert Syndrome
* Known sensitivities to toxins
* Severe bradycardia (HR<50 bpm) or hypotension (systolic blood pressure of <80 mmHg)
* Deep vein thrombosis treatment doses of anticoagulants or coumadin
* History of recent dysphagia
* Ventilator dependent
* Unstable cervical fracture or not surgically stabilized

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Maerz, MD, Principal Investigator — Craig Hospital
Locations (1):
- Craig Hospital, Englewood, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants that met eligibility criteria were enrolled from April 2006 through August 2008. All participants were enrolled while undergoing inpatient rehabilitation at Craig Hospital. 19 individuals were enrolled and randomized into the study.
Groups:
- Group 1-Botox A Group: This group received the active drug, botox a injections.
- Group 2-saline Group: Group 2 is the control group and received injections of saline instead of the saline plus botox A injections that the treatment group received
Period: Overall Study
Arm/Group | Group 1-Botox A Group | Group 2-saline Group
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1-Botox A Group | Group 2-saline Group | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (14.44) | 35.91 (11) | 36.15 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Scale-NRS
Description: The Numerical Rating Scale (NRS) is a numerical scale from 0-10 used to rate pain. Participants were asked to assess the worst pain experienced in the past 5 days and rate it on a numerical scale from 0-10, with 10 being the "worst possible pain" they have experienced and 0 being "no pain."
Time Frame: 6 weeks post-injection
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Group 1-Botox A Group: Those randomized to this treatment group received injections based on treatment plan designed by PI and study physical therapist. Botulism toxin A was diluted in 25 cc of saline for the injections. Multiple injections may have occured during a single clinic visit based on pain/stiffness upon assesment by the study treatment team.
- Group 2-saline Group: Those randomized to this treatment group received injections based on treatment plan devised by study PI and study physical therapist. 25 cc of saline were used for these injections. Multiple injections may have occured during a single clinic visit based on pain/stiffness upon assesment by the study treatment team.
Arm/Group | Group 1-Botox A Group | Group 2-saline Group
Number analyzed (Participants) | 10 | 9
units on a scale | 4.50 [2.58 to 6.42] | 3.44 [1.42 to 5.46]
Statistical Analysis 1: Comparison: Group 1-Botox A Group vs Group 2-saline Group; Test type: Superiority or Other; p = 0.432, ANCOVA

2. Secondary Outcome: Brief Pain Inventory-Short Form - Interference Score
Description: Interference in daily activities was measured with the Brief Pain Inventory (BPI) Interference Score. Participants rated the extent to which pain interfered with their participation in six general activities during the past week, using a scale of 0 (does not interfere) to 10 (completely interferes). Note that for the purposes of this study, the question regarding walking was removed from the original scale which has seven items). Mean score across the 6 items was calculated (range could be 0 - 10) with higher score indicating more pain interference.
Time Frame: 6 months post-injection
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Group 1 - Botox A | Group 2 - Saline Group
Number analyzed (Participants) | 10 | 9
units on a scale | 3.19 [1.65 to 4.73] | 1.62 [0.08 to 3.16]

ADVERSE EVENTS:
Arm/Group | Group 1-Botox A Group | Group 2-saline Group
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9

LIMITATIONS AND CAVEATS:
Study outcome measures modified to reflect available study results. AE's monitored daily; specific data is not available (study completed >10yrs ago). Investigator summary indicates no SAE's/AE's related to study intervention (treatment or sham).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No